CLINICAL TRIAL: NCT04574908
Title: A Pilot Trial of Continuous Portable Postoperative Hemodynamic And Saturation Monitoring On Hospital Wards
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00063530
Record Dates: First submitted 2020-09-28; First posted 2020-10-05 (Actual); Results first posted 2022-11-22 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2021-10

CONDITIONS: Hemodynamic Instability; Respiratory Complications of Care
Keywords: postoperative care; postoperative monitoring; vital signs; portable monitor

STUDY DESIGN:
Who Masked: Participant
Masking Description: The 2 wards will alternate every 4 weeks as to blinded/unblinded allocations. Blinded will be continuous ward monitoring with alarms silenced and screens covered; unblinded will be continuous monitoring accessible to clinicians with pre-specified alerts at MAP <65 mmHg, heart rate >110 b/m, and SpO2 <90%. Of note, to ensure patient safety and no risk in either arm, factory alarm limits (see table under human subjects protection) at extremes of physiological vital signs will stay on in the blinded/silenced arm, and both arms will have every 4 hourly checks by nursing teams.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Blinded Ward (Active Comparator): Continuous ward monitoring with hallway monitor screens covered. When an alarm goes off (limits based on the stratification of that month) the nursing staff will still be notified via their Ascom phone as per standard of care. Nursing staff will log in to WakeOne to verify the vital sign and/or go to the patient room to check on the patient. To ensure patient safety, factory alarm limits at extremes of physiological vital signs will stay on in the blinded arm. Every 4 hourly checks by nursing teams unless otherwise ordered.Continuous monitoring accessible to clinicians with pre-specified alerts at Systolic Blood Pressure alert <70, no Mean Arterial Pressure alert, heart rate >150 beats per minute (b/m), and peripheral capillary oxygen saturation (SpO2) <80%. Every 4 hourly checks by nursing teams unless otherwise ordered. These alarms are consistent with current standard of care.
  Interventions: Device: ViSi device
- Unblinded Ward (Experimental): Continuous ward monitoring with hallway monitor screens accessible for viewing but with alarm limits more narrow. When an alarm goes off (limits based on the stratification of that month) the nursing staff will still be notified via their Ascom phone as per standard of care. Nursing staff will be able to view the hallway monitors showing the vital signs in all of the rooms and/or log in to WakeOne to verify the vital sign and/or go to the patient room to check on the patient. To ensure patient safety, factory alarm limits at extremes of physiological vital signs will stay on in the blinded arm. Every 4 hourly checks by nursing teams unless otherwise ordered. Continuous monitoring accessible to clinicians with pre-specified alerts at Mean Arterial Pressure (MAP) <65 mmHg, heart rate >110 beats per minute (b/m), and peripheral capillary oxygen saturation (SpO2) <90%. Every 4 hourly checks by nursing teams unless otherwise ordered.
  Interventions: Device: ViSi device

INTERVENTIONS:
Device: ViSi device — Mobile patient monitoring system for vital signs.

SUMMARY:
The study team will collect data for this study from participants who are having surgery and recovering postoperatively on 2 pre-designated hospital units. The study team will use vital signs data from a portable device that participants wear on their wrists as well as conventional vital signs data that is collected when a health care provider comes into their room and collect this information.

A substudy is also being performed with the distribution of surveys to the nursing staff on the floors who are utilizing the ViSi hemodynamic monitors within our institution.

DETAILED DESCRIPTION:
This proposed study will provide the necessary preliminary data for a National Institutes of Health Research Grant Project (NIH R01) application that will test the utility of continuous portable hemodynamic monitoring in a large-scale randomized trial. Two separate post surgical hospital units will be randomized to utilize the Sotera ViSi monitoring system or to not utilize the Sotera ViSi monitoring system for a 4 week period of time alternating over the period of 1 year. The study team will assess the effect of unblinded continuous monitoring and the associated alerts on the cumulative duration (min/hour) of each of hypotension, tachycardia, and desaturation. The study team will assess the effect of continuous monitoring and associated alerts on the ordinal clinical intervention outcome which measures the single most extreme/elevated clinical intervention incurred by a patient for any of the 3 outcome variables of interest (hypotension, tachycardia, hypoxia) during the study period with response by staff. The study team will assess the treatment effect on myocardial injury after non-cardiac surgery (MINS) during the study period.

A substudy involving the the medical center nursing staffs' impressions of the device as well as their confidence in its utilization in keeping their assigned patient's safe will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* >/= 65 years of age
* >/= 45 years of age with at least 1 cardiovascular risk (hypertension, diabetes)
* Requiring a general or regional anesthetic as part of their surgical procedure.
* Requiring (or anticipated to require) at least a 48 hour hospital stay after surgery.
* All subjects aged 18 and older who are patients receiving ViSi monitoring on the 2 nursing units involved.

Exclusion Criteria:

* < 48 hour hospital stay
* Receiving local anesthetic for their surgical procedure
* troponins not ordered if <65 years of age without a single cardiovascular risk factor or <45 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 879 (Actual)
Dates: Start 2020-10-07 (Actual); Primary Completion 2021-10-06 (Actual); Study Completion 2021-10-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ashish Khanna, M.D., Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest Univesity Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the IPD collected during the course of the study will be deidentified and then analyzed
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: immediately following publication. No end date available.
Access Criteria: any purpose

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Blinded Ward | Unblinded Ward
Started | 431 | 448
Completed | 431 | 448
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Blinded Ward | Unblinded Ward | Total
Number analyzed (Participants) | 431 | 448 | 879
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 71.16 [63.39 to 80.15] | 70.65 [62.63 to 78.00] | 70.74 [63.20 to 78.78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 236 | 247 | 483
  Male | 195 | 201 | 396
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 3 | 4
  Asian | 3 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 68 | 73 | 141
  White | 348 | 360 | 708
  More than one race | 10 | 11 | 21
  Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Duration of Hypotension in Minutes
Description: Hypotension defined as MAP <65 mmHg.
Time Frame: Ward Admission Through 3rd Postoperative Morning or 48 Continuous Hours (Whichever Comes Earlier)
Measure: Median (Inter-Quartile Range); unit: Minutes
Arm/Group | Blinded Ward | Unblinded Ward
Number analyzed (Participants) | 431 | 448
Minutes | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00]

2. Primary Outcome: Duration of Tachycardia in Minutes
Description: Tachycardia defined as >110 beats/min.
Time Frame: Ward Admission Through 3rd Postoperative Morning or 48 Continuous Hours (Whichever Comes Earlier)
Measure: Median (Inter-Quartile Range); unit: Minutes
Arm/Group | Blinded Ward | Unblinded Ward
Number analyzed (Participants) | 431 | 448
Minutes | 0.01 [0.00 to 0.04] | 0.01 [0.00 to 0.04]

3. Primary Outcome: Duration of Hypoxemia (SpO2 < 90%) in Minutes
Description: Duration of Hypoxemia defined as SpO2 < 90% in Minutes
Time Frame: Ward Admission Through 3rd Postoperative Morning or 48 Continuous Hours (Whichever Comes Earlier)
Measure: Median (Inter-Quartile Range); unit: Minutes
Arm/Group | Blinded Ward | Unblinded Ward
Number analyzed (Participants) | 431 | 448
Minutes | 0.04 [0.01 to 0.09] | 0.03 [0.01 to 0.05]

4. Secondary Outcome: Clinical Nursing Intervention Responses Scale
Description: Clinical nursing intervention responses over the duration of the trial will be categorized as (1) none, (2) independent nursing intervention, (3) notification of physician team, or (4) activation of the hospital Emergency or Rapid Response System. Scale ranges from 1-4 with 4 denoting a worse outcome.
Time Frame: Ward Admission Ward Admission Through 3rd Postoperative Morning or 48 Continuous Hours (Whichever Comes Earlier)
Population: nurses did not enter timely responses in the EMR and therefore there is no data for that outcome measure.
Arm/Group | Blinded Ward | Unblinded Ward
Number analyzed (Participants) | 0 | 0

5. Other Pre Specified Outcome: Incidence of Myocardial Injury After Non-Cardiac Surgery (MINS)
Description: Determined by blood troponin levels. Concentrations ≥0.03 ng/ml will be considered MINS if there is no evidence of a non-ischemic etiology.
Time Frame: Ward Admission Ward Admission Through 3rd Postoperative Morning or 48 Continuous Hours (Whichever Comes Earlier)
Measure: Count of Participants; unit: Participants
Arm/Group | Blinded Ward | Unblinded Ward
Number analyzed (Participants) | 431 | 448
Participants
  yes | 71 | 71
  no | 360 | 377

6. Other Pre Specified Outcome: Patient Satisfaction Survey
Description: Score ranges from 5-50 with higher score denoting better outcome.
Time Frame: Ward discharge on 3rd Postoperative Morning or 48 Continuous Hours (Whichever Comes Earlier)
Population: OM Data not collected
Arm/Group | Blinded Ward | Unblinded Ward
Number analyzed (Participants) | 0 | 0

7. Other Pre Specified Outcome: ViSi Monitor Nursing Staff Survey
Description: Survey showing the nursing perceptions of Certification for Neurophysiological Intraoperative Monitoring (CNIM) as well as the value of these devices in the care of their patients. Survey will obtain impressions of device from nurses. And descriptive statistics will be obtained regarding nurse's impressions of this technology after its having been implemented. Data will be reported via percentages the responses received.
Time Frame: After discharge over a period of 7 days
Population: OM Data not collected
Arm/Group | Blinded Ward | Unblinded Ward
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Hour 72
Arm/Group | Blinded Ward | Unblinded Ward
All-Cause Mortality (participants affected / at risk) | 7/431 | 4/448
Serious Adverse Events (participants affected / at risk) | 7/431 | 4/448
Other Adverse Events (participants affected / at risk) | 0/431 | 0/448
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Blinded Ward (N=431) | Unblinded Ward (N=448)
Death (Cardiac disorders) | 7 (7) | 4 (4) — In Hospital Mortality
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Blinded Ward (N=431) | Unblinded Ward (N=448)
Death (Cardiac disorders) | NA | NA — In Hospital Mortality

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-07-08): https://cdn.clinicaltrials.gov/large-docs/08/NCT04574908/Prot_SAP_002.pdf
  • Informed Consent Form (2021-07-01): https://cdn.clinicaltrials.gov/large-docs/08/NCT04574908/ICF_000.pdf